CLINICAL TRIAL: NCT05579587
Title: Transoral Incisionless Fundoplication (TIF) for Laryngopharyngeal Reflux (LPR) Patients
Acronym: TIF-LPR
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decided not to fund the study.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: EndoGastric Solutions (Industry)
Responsible Party: Principal Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Other Study IDs: 2022P000144
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Laryngopharyngeal Reflux (LPR); Reflux Disease, Gastro-Esophageal; Motility Disorder
Keywords: Transoral Incisionless Fundoplication (TIF); Fundoplication; Nissen Fundoplication; Proton Pump Inhibitor; Esophageal Manometry; Laryngoscopy; HEMII-pH; Reflux Symptom Index (RSI); GERD-HRQL
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- LPR Patients: Adults with a confirmed diagnosis of LPR with HEMII-pH (≥2 LPR events in 24 hr period), Esophageal manometry and Laryngoscopy undergoing endoscopic transoral incisionless fundoplication (TIF).
  Interventions: Device: Transoral Incisionless Fundoplication

INTERVENTIONS:
Device: Transoral Incisionless Fundoplication — Transoral incisionless fundoplication (TIF) is a minimally invasive, endoscopic fundoplication technique. Transoral Incisionless Fundoplication (TIF) is an FDA approved endoluminal fundoplication technique which utilizes EsophyX device to restore the valve at the gastroesophageal junction. The EsophyX device (EndoGastric Solutions, Redmond, Wash, USA) is an FDA approved procedure for chronic of refractory GERD.
  Other Names: TIF

SUMMARY:
In this research study the investigators want to learn more about the effectiveness of an endoscopic procedure (an endoscope is a lighted tube that is placed down the participants esophagus, through the participants mouth) which uses a device that allows the doctor to repair or recreate the body's natural barrier to reflux. It uses preloaded forceps (tweezers) and fasteners and requires no incision to tighten the connection between the participants esophagus and stomach. This procedure is performed to aid in the treatment of symptoms of Gastroesophageal Reflux disease (GERD) in patients with diagnosed Laryngopharyngeal reflux (LPR). LPR is a condition resulting from backflow of stomach contents into the laryngopharynx (connection point in the participants throat through which food, water, and air pass) resulting in symptoms that can be referred to larynx/hypopharynx. The device the investigators will use to perform the transoral incisionless fundoplication procedure (TIF) is called the EsophyX device. The participants have been asked to participate because they have been diagnosed with LPR and have either failed medical therapy (taking prescription proton pump inhibitors (PPI) to reduce stomach acid production or do not want to be on long-term medical treatment.

DETAILED DESCRIPTION:
To date, more than one-third of the motility patients that the investigators see in practice at Brigham and Women's Hospital have LPR. There is currently limited literature available addressing LPR as a primary indication for the TIF procedure moreover there is no single therapy that has proved its efficacy over the years against LPR. The investigators propose a pilot study to investigate the efficacy of TIF with the EsophyX device (EndoGastric Solutions, Inc., Redmond WA, USA) in patients with LPR. The study design would include up to 25 patients to receive the TIF procedure and will take 12 months to complete it. The investigators will compare objective and subjective outcomes at baseline and 3 months post TIF procedure to assess its efficacy against LPR. The investigators will submit the proposal to EndoGastric solutions, anticipating that they will cover part of the funding required to conduct our Pilot Study.

In conclusion, LPR lacks an effective therapy despite posing a significant healthcare burden. Medical therapy with PPI has a variable response, and more invasive Laparoscopic fundoplication is associated with a high risk of unwanted long-term side effects. TIF can potentially bridge this gap between medical and more invasive approaches for the patient population suffering from this condition. It has the potential to prove to be a less invasive and safe treatment indication for patients with chronic or refractory LPR who have either failed medical therapy or do not want to be on long-term medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any adult with a confirmed diagnosis of LPR with HEMII-pH (≥2 LPR events in 24 hr period), Esophageal manometry and Laryngoscopy.
* Having daily bothersome symptoms of LPR.
* Willing and able to cognitively sign a consent form for Surgical treatment of LPR with the TIF.
* Willing and available for follow up visit and repeat testing (HEMII-pH, Esophageal manometry and laryngoscopy) at 3 months post procedure.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unable or unwilling to comply with study procedures
* Body Mass Index >35.
* Hiatal hernia>2cm in axial height and >2cm in greatest transverse dimension.
* Esophagitis grade C and D
* Barrett's esophagus>2cm
* Esophageal ulcer
* Fixed esophageal stricture or narrowing
* Portal hypertension and/or varices
* Active gastro-duodenal ulcer disease; Gastric outlet obstruction or stenosis
* Gastroparesis
* Coagulation disorders
* History of any of the following: resective gastric or esophageal surgery, anti-reflux surgery with anatomy unsuitable for TIF procedure per physician judgment, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis
* Pregnancy or plans of pregnancy in the next 12 months
* Enrollment in another device or drug study that may confound the results.
* Acute or chronic illness or history of illness which in the opinion of the investigator could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data, such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes (HbA1c >12%), etc.
* Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosed Laryngopharyngeal reflux (LPR) who are scheduled for endoscopic transoral incisionless fundoplication procedure (TIF).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
LPR Symptoms | Baseline and 3 months post-procedure
  Number of participants reporting LPR symptom elimination or clinically significant improvement evaluated by RSI (Reflux Symptom Index) and GERD-HRQL Questionnaire.
LPR Events | Baseline and 3 months post-procedure
  Number of participants with reduced LPR events as evaluated by HEMII-pH

SECONDARY OUTCOMES:
GERD Symptoms | Baseline and 3 months post-procedure
  Elimination of Daily bothersome GERD symptoms evaluated by GERD-HRQL Questionnaire
Patient Satisfaction | Baseline and 3 months post-procedure
  Patients Satisfaction evaluated by GERD-HRQL Questionnaire
Lower Esophageal Sphincter Tone | Baseline and 3 months post-procedure
  Change in Lower esophageal sphincter tone evaluated by Esophageal manometry
Laryngopharyngeal anatomy | Baseline and 3 months post-procedure
  Change in Laryngopharyngeal anatomy evaluated by Laryngoscopy
PPI Discontinuation | Baseline and 3 months post-procedure
  Discontinuation of PPI's

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share data will be on a case by case basis. The other researchers may contact the PI and discuss study plans. An agreement through Mass General Brigham will need to be executed prior to sharing the de-identified data.

REFERENCES:
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Background] Koufman JA. The otolaryngologic manifestations of gastroesophageal reflux disease (GERD): a clinical investigation of 225 patients using ambulatory 24-hour pH monitoring and an experimental investigation of the role of acid and pepsin in the development of laryngeal injury. Laryngoscope. 1991 Apr;101(4 Pt 2 Suppl 53):1-78. doi: 10.1002/lary.1991.101.s53.1. PMID 1895864
- [Background] Francis DO, Rymer JA, Slaughter JC, Choksi Y, Jiramongkolchai P, Ogbeide E, Tran C, Goutte M, Garrett CG, Hagaman D, Vaezi MF. High economic burden of caring for patients with suspected extraesophageal reflux. Am J Gastroenterol. 2013 Jun;108(6):905-11. doi: 10.1038/ajg.2013.69. Epub 2013 Apr 2. PMID 23545710
- [Background] Spantideas N, Drosou E, Bougea A, AlAbdulwahed R. Proton Pump Inhibitors for the Treatment of Laryngopharyngeal Reflux. A Systematic Review. J Voice. 2020 Nov;34(6):918-929. doi: 10.1016/j.jvoice.2019.05.005. Epub 2019 May 31. PMID 31160182
- [Background] Fraser LA, Leslie WD, Targownik LE, Papaioannou A, Adachi JD; CaMos Research Group. The effect of proton pump inhibitors on fracture risk: report from the Canadian Multicenter Osteoporosis Study. Osteoporos Int. 2013 Apr;24(4):1161-8. doi: 10.1007/s00198-012-2112-9. Epub 2012 Aug 14. PMID 22890365
- [Background] Lazarus B, Chen Y, Wilson FP, Sang Y, Chang AR, Coresh J, Grams ME. Proton Pump Inhibitor Use and the Risk of Chronic Kidney Disease. JAMA Intern Med. 2016 Feb;176(2):238-46. doi: 10.1001/jamainternmed.2015.7193. PMID 26752337
- [Background] Ciovica R, Gadenstatter M, Klingler A, Lechner W, Riedl O, Schwab GP. Quality of life in GERD patients: medical treatment versus antireflux surgery. J Gastrointest Surg. 2006 Jul-Aug;10(7):934-9. doi: 10.1016/j.gassur.2006.04.001. PMID 16843863
- [Background] Galmiche JP, Hatlebakk J, Attwood S, Ell C, Fiocca R, Eklund S, Langstrom G, Lind T, Lundell L; LOTUS Trial Collaborators. Laparoscopic antireflux surgery vs esomeprazole treatment for chronic GERD: the LOTUS randomized clinical trial. JAMA. 2011 May 18;305(19):1969-77. doi: 10.1001/jama.2011.626. PMID 21586712
- [Background] McCarty TR, Itidiare M, Njei B, Rustagi T. Efficacy of transoral incisionless fundoplication for refractory gastroesophageal reflux disease: a systematic review and meta-analysis. Endoscopy. 2018 Jul;50(7):708-725. doi: 10.1055/a-0576-6589. Epub 2018 Apr 6. PMID 29625507
- [Background] Testoni S, Hassan C, Mazzoleni G, Antonelli G, Fanti L, Passaretti S, Correale L, Cavestro GM, Testoni PA. Long-term outcomes of transoral incisionless fundoplication for gastro-esophageal reflux disease: systematic-review and meta-analysis. Endosc Int Open. 2021 Feb;9(2):E239-E246. doi: 10.1055/a-1322-2209. Epub 2021 Feb 3. PMID 33553587
- [Background] Barnes WE, Hoddinott KM, Mundy S, Williams M. Transoral incisionless fundoplication offers high patient satisfaction and relief of therapy-resistant typical and atypical symptoms of GERD in community practice. Surg Innov. 2011 Jun;18(2):119-29. doi: 10.1177/1553350610392067. Epub 2011 Feb 8. PMID 21307014
- [Background] Wilson EB, Barnes WE, Mavrelis PG, Carter BJ, Bell RC, Sewell RW, Ihde GM, Dargis D, Hoddinott KM, Shughoury AB, Gill BD, Fox MA, Turgeon DG, Freeman KD, Gunsberger T, Hausmann MG, Leblanc KA, Deljkich E, Trad KS. The effects of transoral incisionless fundoplication on chronic GERD patients: 12-month prospective multicenter experience. Surg Laparosc Endosc Percutan Tech. 2014 Feb;24(1):36-46. doi: 10.1097/SLE.0b013e3182a2b05c. PMID 24487156
- [Background] Trad KS, Barnes WE, Prevou ER, Simoni G, Steffen JA, Shughoury AB, Raza M, Heise JA, Fox MA, Mavrelis PG. The TEMPO Trial at 5 Years: Transoral Fundoplication (TIF 2.0) Is Safe, Durable, and Cost-effective. Surg Innov. 2018 Apr;25(2):149-157. doi: 10.1177/1553350618755214. Epub 2018 Feb 6. PMID 29405886
- [Background] Borges LF, Chan WW, Carroll TL. Dual pH Probes Without Proximal Esophageal and Pharyngeal Impedance May Be Deficient in Diagnosing LPR. J Voice. 2019 Sep;33(5):697-703. doi: 10.1016/j.jvoice.2018.03.008. Epub 2018 Aug 3. PMID 30082108
- [Background] Carroll TL, Nahikian K, Asban A, Wiener D. Nissen Fundoplication for Laryngopharyngeal Reflux After Patient Selection Using Dual pH, Full Column Impedance Testing: A Pilot Study. Ann Otol Rhinol Laryngol. 2016 Sep;125(9):722-8. doi: 10.1177/0003489416649974. Epub 2016 May 23. PMID 27217426
- [Background] Hoppo T, Komatsu Y, Jobe BA. Antireflux surgery in patients with chronic cough and abnormal proximal exposure as measured by hypopharyngeal multichannel intraluminal impedance. JAMA Surg. 2013 Jul;148(7):608-15. doi: 10.1001/jamasurg.2013.1376. PMID 23700139
- [Background] Zerbib F, Roman S, Bruley Des Varannes S, Gourcerol G, Coffin B, Ropert A, Lepicard P, Mion F; Groupe Francais De Neuro-Gastroenterologie. Normal values of pharyngeal and esophageal 24-hour pH impedance in individuals on and off therapy and interobserver reproducibility. Clin Gastroenterol Hepatol. 2013 Apr;11(4):366-72. doi: 10.1016/j.cgh.2012.10.041. Epub 2012 Nov 8. PMID 23142603
- See also: Safety information for the TIF procedure — https://www.endogastricsolutions.com/technology/safety-info/